CLINICAL TRIAL: NCT00404677
Title: The Correlation Between Airway Inflammation and Loss of Deep Inhalation Bronchoprotection in Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Dr. Don Cockcroft, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BIO-REB 06-92; BIO-REB 06-92
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (2):
- Standard (Placebo Comparator): Methacholine challenges are performed using the standardized two minute tidal breathing method
  Interventions: Other: deep inhalation
- Modified (Active Comparator): Five deep inhalation maneouvers are incorporated into the standardized methacholine challenge
  Interventions: Other: deep inhalation

INTERVENTIONS:
Other: deep inhalation — deep inhalation is comprised of an inhalation manoeuver from FRC to TLC

SUMMARY:
The loss of deep inhalation bronchoprotection in asthmatic individuals has been shown to be related to the degree of airway hyperresponsiveness, a hallmark of asthma. In several studies, asthmatic individuals with mild airway hyperresponsiveness (AHR) (methacholine PC20 > 2 mg/mL) had a difference in methacholine PC20 with and without deep inhalations that averaged 1.8 doubling methacholine concentrations (p=0.0003). Conversely, asthmatic individuals with moderate to severe AHR (methacholine PC20 ≤ 2 mg/mL) had a non-significant difference in methacholine PC20 with and without deep inhalations (p=0.09). This loss of deep inhalation bronchoprotection is also now believed to play an important role in the pathogenesis of asthma. Airway inflammation is another of the key features of asthma and information on airway inflammation is increasingly being used in the diagnosis and treatment of asthma. The level of airway inflammation (as measured by fraction of exhaled nitric oxide and sputum eosinophilia) has also been shown to be correlated to the level of airway hyperresponsiveness (as measured by methacholine PC20). In addition, glucocorticoids have been shown to decrease airway hyperresponsiveness, further suggesting that these two phenomena, airway inflammation and airway hyperresponsiveness, are related. We therefore suggest that the degree of airway inflammation is related to the loss of deep inhalation bronchoprotection and expect there to be a negative correlation between the degree of deep inhalation bronchoprotection and airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of asthma

Exclusion Criteria:

* other lung disease(s)
* smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
fraction of exhaled nitric oxide, sputum eosinophils and methacholine PC20 | freaction of exhaled nitric oxide data collected prior to methacholine challenges; sputum collected after the first methacholine challenge

CONTACTS AND LOCATIONS:
Overall Officials: Donald Cockcroft, MD, FRCP(C), Principal Investigator — Department of Medicine, Division of Respirology, Critical Care and Sleep Medicine, University of Saskatchewan